CLINICAL TRIAL: NCT06351124
Title: Feasibility of Beta-hydroxybutyrate Supplementation to Reduce Inflammation in Patients with Inflammatory Bowel Disease
Brief Title: Beta-Hydroxybutyrate Feasibility Treating IBD
Acronym: BHB
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00005294
Record Dates: First submitted 2024-03-26; First posted 2024-04-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Crohn's Disease; Inflammatory Bowel Diseases
Keywords: Beta-hydroxybutyrate (BHB); proinflammatory immune cells; gut bacteria; ketone body; ketogenesis; gut barrier integrity; inflammation; digestive health
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: This will be a prospective, open-label, randomized, two-arm pilot trial of adults
Masking Description: Eligible consenting patients will be randomized to either standard of care therapy (control) vs standard of care therapy plus BHB supplementation (intervention). BHB will be supplemented as a capsule taken orally three times daily for four weeks for those randomized to the intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard of care therapy (control) (No Intervention): Arm does not receive the BHB supplement
- Standard of care therapy plus BHB supplementation (intervention). (Active Comparator): Arm does receives the BHB supplement
  Interventions: Biological: Feasibility of beta-hydroxybutyrate supplementation to reduce inflammation in patients with Crohn's

INTERVENTIONS:
Biological: Feasibility of beta-hydroxybutyrate supplementation to reduce inflammation in patients with Crohn's — Is Beta-hydroxybutyrate a supplement that can control symptoms and progression of Crohn's.
  Other Names: BHB Feasibility
  Arms: Standard of care therapy plus BHB supplementation (intervention).

SUMMARY:
This clinical trial aims to understand the feasibility of patients taking ketone body supplement beta-hydroxybutyrate (BHB) for 4 weeks with a confirmed diagnosis of Crohn's disease and starting new therapy for active disease.

The main questions it aims to answer are:

* BHB supplementation will be feasible and acceptable to patients.
* BHB supplementation will be associated with a reduction in systemic inflammation.
* BHB supplementation will be associated with a reduction in pro-inflammatory bacterial colonies.

Participants will:

* Take 3 capsules x 3 times per day for 4 weeks.
* Document food consumption using a 24-hour food recall questionnaire.
* Provide blood and fecal samples twice, at the beginning of the study and the 4-week mark.

Researchers will compare the group taking the ketone body supplement and the group not taking the supplement to see if the supplement provides relief of symptoms suffered from Crohn's disease.

DETAILED DESCRIPTION:
A clinical trial designed to determine the feasibility of prebiotic supplementation with beta-hydroxybutyrate (BHB) in Crohn's patients in a prospective, open-label pilot trial and to assess the association between BHB supplementation and changes in the microbiome, inflammation, and markers of disease severity in Crohn's patients in a prospective pre-/post-study design.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Confirmed diagnosis of Crohn's disease
* Active disease defined as either a fecal calprotectin >250 µg/g or active disease on endoscopy within the prior 3 months
* Starting a new therapy defined as a biologic (anti-TNF, anti-integrin, IL-12/23, or IL-23) or small molecule therapy (JAK inhibitor, S1P receptor modulator)
* Willing to provide consent for participation.
* Managed at UT Digestive Health Clinic.

Exclusion Criteria:

* Any current or recent (within 4 weeks) use of BHB supplement
* Currently or recently (within 4 weeks) following a ketogenic diet
* Currently or recently (within 4 weeks) following an intermittent fasting diet
* Any recent antibiotic use (within 3 months)
* Recent infection with C. difficile (within 6 months)
* Current or recent (within 4 weeks) daily use of acid-suppressing therapy (proton pump inhibitor or H2 receptor blocker)
* Current or recent use (within four weeks) of non-dietary probiotic supplements
* Unwilling to provide signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ability to enroll patients who meet the inclusion criteria within the target time frame | 12 months
  Number of patients recruited
Adherence to proposed study timelines and anticipated study costs | 12 months
  Alignment of predicted timeline and costs to real timeline and costs
Patient adherence to the intervention | 12 months
  How many dosages do participants miss following the regiment.

SECONDARY OUTCOMES:
Microbial Diversity | 4 weeks
  Changes in the microbial diversity and proportional abundance of major bacterial taxa at four weeks compared to baseline
BHB Blood Levels | 4 weeks
  Changes in BHB serum levels at baseline compared to 4 weeks
Gastrointestinal Symptoms | 4 weeks
  Changes in (GI PROMIS score)
Pain intensity (Patient-Reported Outcomes Measurement Information System (PROMIS) | 4 weeks
  Changes in (PROMIS-29), PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain.
  Scales:
  Physical Function 5-1: 5.without any difficulty, 4.with a little difficulty, 3.with some difficulty, 2.with much difficulty, 1.unable Anxiety & Depression 1-5: 1.Never, 2.Rarely, 3.Sometimes, 4.Often, 5.Always Fatigue 5-1: 1.Not at all, 2.A little bit, 3.Somewhat, 2.Quite a bit, 1.Very much Sleep Disturbance 5-1: 5.Very poor, 4.poor 3. fair, 2.Good, 1. very good Ability to participate in social roles and activities 5-1: 5.Never, 4.Rarely, 3.Sometimes, 2.Usually, 1.Always Pain interference 1-5: 1. Not at all, 2.A little bit, 3.Somewhat, 4.Quite a bit, 5.Very much
Clinical Response | 4 weeks
  Improved disease activity (reduction in fecal calprotectin by 50%)
Systemic Inflammation | 4 weeks
  changes measured by C-reactive protein
Adverse Events | 4 weeks
  Adverse events related to the intervention. Outcomes will be assessed at four weeks follow-up
Assess disease activity by Intestinal Ultrasound (IUS) | 4 weeks
  Assess disease activity in patients with inflammatory bowel disease using Intestinal ultrasound (IUS), a noninvasive tool. This can be performed in the clinic at the bedside without any bowel preparation, fasting, or sedation. It is highly acceptable to patients with minimal risk.

CONTACTS AND LOCATIONS:
Overall Officials: Linda A. Feagins, Associate Professor, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No